CLINICAL TRIAL: NCT01544582
Title: An Observational Post-Authorization Safety Study (PASS) of Victrelis™ (Boceprevir) Among Chronic Hepatitis C Patients
Brief Title: Drug Utilization of Boceprevir and Clinical Management of Health Outcomes of Interest in Chronic Hepatitis C Participants (P08518)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P08518; EP08043.001 (Other: Merck Epidemiology Number); SCH 503034 P08518 (Other: Schering Protocol Number); MK-3034-072 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-02-02; First posted 2012-03-06 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C Chronic
Keywords: Pegylated Interferon; boceprevir; telaprevir
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Boceprevir + PR: CHC genotype-1 participants included in study and prescribed boceprevir plus PR as routine clinical management.
- Telaprevir + PR: CHC genotype-1 participants included in study and prescribed telaprevir plus PR as routine clinical management.
- PR Alone: CHC genotype-1 participants included in study and prescribed PR alone as routine clinical management.

SUMMARY:
This is an observational prospective follow-up study to assess the utilization of boceprevir and the management of pre-specified health outcomes of interest (HOIs) under conditions of routine clinical care in participants with chronic hepatitis C (CHC) genotype 1.

As an observational prospective study, this study is not intended to change the participant/physician relationship, nor influence the physician's drug prescription or therapeutic management of the participant. No individual administration of any therapeutic or prophylactic agent is assigned in this protocol, and there are no procedures required as part of this protocol. Physician choice of the drug used to treat the participant is based on clinical judgment alone.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic hepatitis C (CHC) genotype-1 infection
* Untreated or failed previous therapy
* Initiated a new treatment regimen after the study implementation date at their site
* Agrees to participate in the study by giving written informed consent

Exclusion Criteria:

* Taking part in a clinical trial or in any study where a participant is receiving care outside of normal clinical practice for Hepatitis C Virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years or older with CHC genotype 1
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 713 Chronic Hepatitis C (CHC) participants included in the study, 679 were included in the Analysis Population and 34 were excluded. The Analysis Population comprised participants receiving Boceprevir plus peginterferon and ribavirin (PR), Telaprevir plus PR, or PR alone.
Groups:
- All Included Participants: All CHC genotype-1 participants included in study.
Period: Screening/Eligibility
Arm/Group | All Included Participants | Boceprevir + PR | Telaprevir + PR | PR Alone
Started | 713 | 0 | 0 | 0
Analysis Population | 679 | 0 | 0 | 0
Completed | 679 (Completed means met criteria for Analysis Population) | 0 | 0 | 0
Not Completed | 34 | 0 | 0 | 0
Not completed — Initiated Different CHC Treatment | 1 | 0 | 0 | 0
Not completed — Eligibility Criteria Not Met | 33 | 0 | 0 | 0
Period: Analysis Population
Arm/Group | All Included Participants | Boceprevir + PR | Telaprevir + PR | PR Alone
Started | 0 (Analysis Population was grouped into Boceprevir+PR, Telaprevir+PR, or PR Alone) | 298 | 307 | 74
Completed | 0 | 180 | 205 | 35
Not Completed | 0 | 118 | 102 | 39
Not completed — Participant Refuses to Continue Study | 0 | 15 | 17 | 4
Not completed — Physician Decision | 0 | 13 | 10 | 9
Not completed — Safety Reason | 0 | 33 | 31 | 8
Not completed — Effectiveness Reason | 0 | 48 | 29 | 12
Not completed — New Contraindication-Alcohol Abuse | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 6 | 6 | 5
Not completed — Bad Tolerance to Treatment | 0 | 0 | 2 | 0
Not completed — Did Not Meet Inclusion Criteria | 0 | 0 | 3 | 0
Not completed — Intolerance | 0 | 1 | 0 | 0
Not completed — Liver Transplantation | 0 | 0 | 1 | 0
Not completed — No Social Insurance | 0 | 0 | 1 | 0
Not completed — Poor Adherence | 0 | 0 | 1 | 0
Not completed — Poor Participant Compliance | 0 | 1 | 0 | 0
Not completed — Programmed Surgery | 0 | 1 | 0 | 0
Not completed — Participant in Jail | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis Population: All CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone | Total
Number analyzed (Participants) | 298 | 307 | 74 | 679
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.3) | 50.1 (10.9) | 46.3 (11.6) | 50.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 102 | 25 | 240
  Male | 185 | 205 | 49 | 439

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone (Drug Utilization Pattern)
Description: The percentage of CHC participants initiating boceprevir plus PR treatment, telaprevir plus PR treatment, or PR treatment alone was determined from a Drug Utilization questionnaire that was administered to physicians using an electronic Case Report Form (eCRF) to collect site level information and reported with 95% confidence intervals.
Time Frame: Up to 37 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Included Participants
Number analyzed (Participants) | 679
percentage of participants
  Initiating Boceprevir + PR Treatment | 43.9 [40.1 to 47.7]
  Initiating Telaprevir + PR Treatment | 45.2 [41.4 to 49.0]
  Initiating PR Treatment Alone | 10.9 [8.7 to 13.5]

2. Primary Outcome: Baseline Characteristics of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone: Weight
Description: Baseline mean weight (standard deviation [SD]) in kilograms (Kg) was recorded from the eCRF.
Time Frame: Before initiation of CHC treatment (Week 0 baseline)
Population: Participants in the Analysis Population (all CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone) with available demographic data (weight).
Measure: Mean (Standard Deviation); unit: kilograms (Kg)
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Number analyzed (Participants) | 280 | 280 | 74
kilograms (Kg) | 77.7 (17.4) | 77.0 (15.5) | 71.7 (13.7)

3. Primary Outcome: Baseline Characteristics of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone: Height
Description: Baseline mean height (SD) in centimeters (cm) was recorded from the eCRF.
Time Frame: Before initiation of CHC treatment (Week 0 baseline)
Population: Participants in the Analysis Population (all CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone) with available demographic data (height).
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Number analyzed (Participants) | 254 | 238 | 61
centimeters | 170.8 (9.8) | 170.8 (8.8) | 171.0 (7.5)

4. Primary Outcome: Baseline Characteristics of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone: Body Mass Index (BMI)
Description: Baseline mean body mass index (SD) in Kg/m^2 was recorded from the eCRF.
Time Frame: Before initiation of CHC treatment (Week 0 baseline)
Population: Participants in the Analysis Population (all CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone) with available demographic data (BMI).
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Number analyzed (Participants) | 248 | 233 | 61
Kg/m^2 | 26.5 (5.1) | 26.5 (4.8) | 24.7 (4.2)

5. Primary Outcome: Baseline Disease Characteristics of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone: Baseline Hepatitis C Virus (HCV) Genotype
Description: Baseline HCV genotype was recorded from the eCRF and the number of participants who were 1a genotype, 1b genotype, or unknown/other was reported.
Time Frame: Before initiation of CHC treatment (Week 0 baseline)
Population: Participants in the Analysis Population (all CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone) with available demographic data (HCV genotype).
Measure: Number; unit: participants
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Number analyzed (Participants) | 298 | 307 | 74
participants
  1a genotype | 107 (5.1) | 120 (4.8) | 33 (4.2)
  1b genotype | 147 | 148 | 30
  Unknown/Other | 44 | 39 | 11

6. Primary Outcome: Baseline Disease Characteristics of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone: Baseline Viral Load
Description: Participant baseline HCV viral load was recorded from the eCRF and categorized as either "Low" (<800,000 IU/mL or <2,000,000 RNA copies/mL) or "High" (≥800,000 IU/mL or ≥2,000,000 RNA copies/mL).
Time Frame: Before initiation of CHC treatment (Week 0 baseline)
Population: Participants in the Analysis Population (all CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone) with available demographic data (viral load).
Measure: Number; unit: participants
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Number analyzed (Participants) | 298 | 307 | 74
participants
  Low (<800,000 IU/mL) | 101 (5.1) | 94 (4.8) | 35 (4.2)
  High (≥800,000 IU/mL) | 182 | 197 | 39
  Unavailable | 15 | 16 | 0

7. Primary Outcome: Baseline Disease Characteristics of Participants Initiating Boceprevir Plus PR Treatment, Telaprevir Plus PR Treatment, or PR Treatment Alone: Baseline Grade for Child-Pugh Score
Description: The Child-Pugh Score is used to determine the prognosis of chronic liver disease, in particular cirrhosis. It is classified into Classes A (best prognosis) to C (worst prognosis). Child-Pugh scores assessed within 3 months before CHC treatment regimen initiation were recorded from the eCRF, and the number of participants who were Grade A, Grade B, Grade C, not assessed, or unknown whether assessed were reported.
Time Frame: Before initiation of CHC treatment (Week 0 baseline)
Population: Participants in the Analysis Population (all CHC genotype-1 participants included in study meeting eligibility criteria and receiving boceprevir plus peginterferon and ribavirin (PR), telaprevir plus PR, or PR alone) with available demographic data (Child Pugh score).
Measure: Number; unit: participants
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Number analyzed (Participants) | 298 | 307 | 74
participants
  Grade A | 97 (5.1) | 61 (4.8) | 30 (4.2)
  Grade B | 1 | 3 | 0
  Grade C | 0 | 0 | 0
  Not Assessed | 169 | 203 | 39
  Unknown whether assessed | 31 | 40 | 5

8. Primary Outcome: Percentage of Anemia Episodes Managed by at Least One Clinical Intervention
Description: Anemia (hemoglobin <10 g/dL) was considered a Health Outcome of Interest (HOI) for this study. Clinical interventions used to manage episodes of anemia in participants could include erythropoiesis stimulating agent (ESA), blood transfusion, drug dose reduction, other treatment, and CHC treatment regimen modifications (drug dose reduction, drug discontinuation, and drug interruption). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive). The percentage of anemia episodes that were managed by at least one intervention is reported for each CHC treatment exposure group with 95% confidence intervals.
Time Frame: Up to 48 weeks of a treatment regimen
Population: Participants in the Analysis Population (all CHC genotype-1 participants included on study meeting eligibility criteria and treated with boceprevir plus PR, telaprevir plus PR, or PR alone) who experienced at least one episode of anemia. Participants categorized by treatment group of exposure (further described in Arm Description).
Measure: Number (95% Confidence Interval); unit: percentage of episodes
Units Other Than Participants: anemia episodes total
Groups:
- PR Group of Exposure: CHC genotype-1 participants included on study who received PR either alone or during the PR lead-in period when combined with boceprevir or telaprevir. For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment group was not mutually exclusive). The PR Treatment Group of Exposure comprised all 74 participants receiving PR only, plus 292 participants from the Boceprevir + PR Treatment Group who received PR during the lead-in period, plus 28 participants from the Telaprevir + PR Treatment Group who received PR during the lead-in period.
- Boceprevir + PR Group of Exposure: CHC genotype-1 participants included on study who received boceprevir + peginterferon and ribavirin (PR) as routine clinical management. For this analysis, participants were categorized by CHC treatment group of exposure. The Boceprevir + PR Treatment Group of Exposure included 298 participants who received boceprevir + PR after the lead-in period to the end of follow-up.
- Telaprevir + PR Group of Exposure: CHC genotype-1 participants included on study who received telaprevir + PR as routine clinical management. For this analysis, participants were categorized by CHC treatment group of exposure. The Telaprevir + PR Treatment Group of Exposure included 307 participants who received telaprevir + PR after the lead-in period to the end of follow-up.
- PR + Boceprevir + Telaprevir Group of Exposure: CHC genotype-1 participants included on study that received telaprevir + PR as routine clinical management and then switched to Boceprevir + PR treatment or vice-versa. For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment group was not mutually exclusive). The PR + Boceprevir+Telaprevir Treatment Group of Exposure included 3 participants who were switched from telaprevir + PR to boceprevir + PR, 2 participants who switched from boceprevir + PR to telaprevir + PR, and one participant who switched from boceprevir + PR to telaprevir + PR, and then to boceprevir + PR during follow-up.
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 27 | 133 | 126 | 4
Number analyzed (anemia episodes total) | 29 | 178 | 166 | 4
percentage of episodes
  % Episodes with ≥1 intervention implemented | 79.3 [60.3 to 92.0] | 72.5 [65.3 to 78.9] | 69.9 [62.3 to 76.7] | 75.0 [19.4 to 99.4]
  % Episodes with no intervention implemented | 20.7 [8.0 to 39.7] | 27.5 [21.1 to 34.7] | 30.1 [23.3 to 37.7] | 25.0 [0.6 to 80.6]

9. Primary Outcome: Percentage of Anemia Episodes Managed by Each Clinical Intervention Out of All Managed Anemia Episodes
Description: Clinical interventions used to manage episodes of anemia in participants could include erythropoiesis stimulating agent (ESA), blood transfusion (BT), other treatment (OT), and CHC treatment regimen modifications including drug dose reduction (DDR), drug discontinuation (DD), and drug interruption (DI). Interventions could be used in combination (e.g. ESA plus blood transfusion) and more than one treatment modification could have been performed. For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive).
  For each CHC treatment exposure group, the percentage of anemia episodes managed by a particular intervention are reported out of the total number of managed anemia episodes with data available for that intervention (i.e. anemia episodes with missing data for an intervention were excluded).
Time Frame: Up to 48 weeks of a treatment regimen
Population: as for outcome 8
Measure: Number; unit: percentage of episodes
Units Other Than Participants: managed anemia episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 27 | 133 | 126 | 4
Number analyzed (managed anemia episodes total) | 23 | 129 | 116 | 3
percentage of episodes
  ESA (managed episodes=21, 124, 114, 3) | 52.4 [60.3 to 92.0] | 46.0 [65.3 to 78.9] | 43.9 [62.3 to 76.7] | 66.7 [19.4 to 99.4]
  BT (managed episodes=21, 125, 115, 3) | 52.4 [8.0 to 39.7] | 20.0 [21.1 to 34.7] | 24.3 [23.3 to 37.7] | 33.3 [0.6 to 80.6]
  OT (managed episodes=22, 127, 115, 3) | 9.1 | 8.7 | 2.6 | 33.3
  DDR (managed episodes=19, 111, 91, 3) | 100.0 | 92.8 | 95.6 | 66.7
  DD (managed episodes=19, 111, 91, 3) | 26.3 | 11.7 | 5.5 | 0.0
  DI (managed episodes=19, 111, 91, 3) | 15.8 | 3.6 | 5.5 | 33.3

10. Primary Outcome: Percentage of Grade 3/4 Neutropenia Episodes Managed by at Least One Clinical Intervention
Description: Grade 3/4 neutropenia (Grade 3: neutrophil count 0.5 - <0.75 × 10^9/L, Grade 4: <0.5 × 10^9/L) was considered a HOI for this study. Clinical interventions used to manage episodes of grade 3/4 neutropenia in participants could include Granulocyte colony-stimulating factor (G-CSF) use and CHC treatment regimen modifications (drug dose reduction, drug discontinuation, and drug interruption). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive). The percentage of grade 3/4 neutropenia episodes that were managed by at least one intervention is reported for each CHC treatment exposure group with 95% confidence intervals.
Time Frame: Up to 48 weeks of a treatment regimen
Population: Participants in the Analysis Population (all CHC genotype-1 participants included on study meeting eligibility criteria and treated with boceprevir plus PR, telaprevir plus PR, or PR alone) who experienced at least one episode of grade 3/4 neutropenia. Participants categorized by treatment group of exposure (further described in Arm Description).
Measure: Number (95% Confidence Interval); unit: percentage of episodes
Units Other Than Participants: Gr 3/4 neutropenia episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 27 | 81 | 46 | 3
Number analyzed (Gr 3/4 neutropenia episodes total) | 30 | 116 | 65 | 3
percentage of episodes
  % Episodes with ≥1 intervention implemented | 36.7 [19.9 to 56.1] | 33.6 [25.1 to 43.0] | 18.5 [9.9 to 30.0] | 0.0 [0.0 to 70.8]
  % Episodes with no intervention implemented | 63.3 [43.9 to 80.1] | 66.4 [57.0 to 74.9] | 81.5 [70.0 to 90.1] | 100.0 [29.2 to 100.0]

11. Primary Outcome: Percentage of Grade 3/4 Neutropenia Episodes Managed by Each Clinical Intervention Out of All Managed Episodes
Description: Clinical interventions used to manage episodes of grade 3/4 neutropenia in participants could include Granulocyte colony-stimulating factor (G-CSF) use, other treatment (OT), and CHC treatment regimen modifications including drug dose reduction (DDR), drug discontinuation (DD), and drug interruption (DI). More than one treatment modification could have been performed. For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive).
  For each CHC treatment exposure group, the percentage of grade 3/4 neutropenia episodes managed by a particular intervention are reported out of the total number of managed grade 3/4 neutropenia episodes with data available for that intervention (i.e. grade 3/4 neutropenia episodes with missing data for an intervention were excluded).
Time Frame: Up to 48 weeks of a treatment regimen
Population: as for outcome 10
Measure: Number; unit: percentage of episodes
Units Other Than Participants: managed neutropenia episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 27 | 81 | 46 | 3
Number analyzed (managed neutropenia episodes total) | 11 | 39 | 12 | 0
percentage of episodes
  G-CSF (managed episodes=11, 39, 12, 0) | 27.3 [19.9 to 56.1] | 46.2 [25.1 to 43.0] | 75.0 [9.9 to 30.0] | NA [0.0 to 70.8] — There were no managed neutropenia episodes in this arm.
  OT (managed episodes=10, 39, 11, 0) | 0.0 [43.9 to 80.1] | 0.0 [57.0 to 74.9] | 0.0 [70.0 to 90.1] | NA [29.2 to 100.0] — There were no managed neutropenia episodes in this arm.
  DDR (managed episodes=8, 24, 5, 0) | 87.5 | 87.5 | 80.0 | NA — There were no managed neutropenia episodes in this arm.
  DD (managed episodes=8, 24, 5, 0) | 25.0 | 12.5 | 0.0 | NA — There were no managed neutropenia episodes in this arm.
  DI (managed episodes=8, 24, 5, 0) | 25.0 | 8.3 | 20.0 | NA — There were no managed neutropenia episodes in this arm.

12. Primary Outcome: Percentage of Grade 3/4 Thrombocytopenia Episodes Managed by at Least One Clinical Intervention
Description: Grade 3/4 thrombocytopenia (Grade 3: platelet count 25 - <50 × 10^9/L, Grade 4: <25 × 10^9/L) was considered a HOI for this study. Clinical interventions used to manage episodes of grade 3/4 thrombocytopenia in participants could include thrombopoietin, platelet transfusion, other treatment, and CHC treatment regimen modifications (drug dose reduction, drug discontinuation, and drug interruption). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive). The percentage of grade 3/4 thrombocytopenia episodes that were managed by at least one intervention is reported for each CHC treatment exposure group with 95% confidence intervals.
Time Frame: Up to 48 weeks of a treatment regimen
Population: Participants in Analysis Population (all CHC genotype-1 participants included on study meeting eligibility criteria and treated with boceprevir plus PR, telaprevir plus PR, or PR alone) who experienced at least one episode of grade 3/4 thrombocytopenia. Participants categorized by treatment group of exposure (further described in Arm Description).
Measure: Number (95% Confidence Interval); unit: percentage of episodes
Units Other Than Participants: Gr 3/4 thrombocytopenia episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 21 | 42 | 37 | 2
Number analyzed (Gr 3/4 thrombocytopenia episodes total) | 26 | 53 | 56 | 2
percentage of episodes
  % Episodes with ≥1 intervention implemented | 42.3 [23.4 to 63.1] | 35.8 [23.1 to 50.2] | 32.1 [20.3 to 46.0] | 0.0 [0.0 to 84.2]
  % Episodes with no intervention implemented | 57.7 [36.9 to 76.6] | 64.2 [49.8 to 76.9] | 67.9 [54.0 to 79.7] | 100.0 [15.8 to 100.0]

13. Primary Outcome: Percentage of Grade 3/4 Thrombocytopenia Episodes Managed by Each Clinical Intervention Out of All Managed Episodes
Description: Clinical interventions used to manage episodes of grade 3/4 thrombocytopenia in participants could include thrombopoietin (TPO), platelet transfusion (PT), other treatment (OT) , and CHC treatment regimen modifications including drug dose reduction (DDR), drug discontinuation (DD), and drug interruption (DI). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive).
  For each CHC treatment exposure group, the percentage of grade 3/4 thrombocytopenia episodes managed by a particular intervention are reported out of the total number of managed grade 3/4 thrombocytopenia episodes with data available for that intervention (i.e. grade 3/4 thrombocytopenia episodes with missing data for an intervention were excluded).
Time Frame: Up to 48 weeks of a treatment regimen
Population: as for outcome 12
Measure: Number; unit: percentage of episodes
Units Other Than Participants: managed thrombocytopenia episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 21 | 42 | 37 | 2
Number analyzed (managed thrombocytopenia episodes total) | 11 | 19 | 18 | 0
percentage of episodes
  TPO (managed episodes=10, 19, 18, 0) | 30.0 [23.4 to 63.1] | 42.1 [23.1 to 50.2] | 11.1 [20.3 to 46.0] | NA [0.0 to 84.2] — There were no managed thrombocytopenia episodes in this arm.
  PT (managed episodes=10, 19, 18, 0) | 0.0 [36.9 to 76.6] | 5.3 [49.8 to 76.9] | 11.1 [54.0 to 79.7] | NA [15.8 to 100.0] — There were no managed thrombocytopenia episodes in this arm.
  OT (managed episodes=9, 17, 18, 0) | 0.0 | 5.9 | 0.0 | NA — There were no managed thrombocytopenia episodes in this arm.
  DDR (managed episodes=11, 10, 15, 0) | 100.0 | 70.0 | 80.0 | NA — There were no managed thrombocytopenia episodes in this arm.
  DD (managed episodes=11, 10, 15, 0) | 18.2 | 20.0 | 26.7 | NA — There were no managed thrombocytopenia episodes in this arm.
  DI (managed episodes=11, 10, 15, 0) | 0.0 | 30.0 | 6.7 | NA — There were no managed thrombocytopenia episodes in this arm.

14. Primary Outcome: Percentage of Serious Rash Episodes Managed by at Least One Clinical Intervention
Description: Serious rash was considered a HOI for this study and included rash > 50% of body surface area, rash associated with significant systemic symptoms, or rash resulting in hospitalization or urgent care visit. Clinical interventions used to manage episodes of serious rash in participants could include topical corticosteroid use, intravenous (IV) and/or oral corticosteroids, emollients/moisturizers, antihistamines, other treatment, and CHC treatment regimen modifications (drug dose reduction, drug discontinuation, and drug interruption). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive). The percentage of serious rash episodes that were managed by at least one intervention is reported for each CHC treatment exposure group with 95% confidence intervals.
Time Frame: Up to 48 weeks of a treatment regimen
Population: Participants in the Analysis Population (all CHC genotype-1 participants included on study meeting eligibility criteria and treated with boceprevir plus PR, telaprevir plus PR, or PR alone) who experienced at least one episode of serious rash. Participants categorized by treatment group of exposure (further described in Arm Description).
Measure: Number (95% Confidence Interval); unit: percentage of episodes
Units Other Than Participants: serious rash episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure
Number analyzed (Participants) | 1 | 7 | 26
Number analyzed (serious rash episodes total) | 1 | 7 | 27
percentage of episodes
  Episodes with ≥1 intervention implemented | 100.0 [2.5 to 100.0] | 100.0 [59.0 to 100.0] | 96.3 [81.0 to 99.9]
  Episodes with no intervention implemented | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 41.0] | 3.7 [0.1 to 19.0]

15. Primary Outcome: Percentage of Serious Rash Episodes Managed by Each Clinical Intervention Out of All Managed Episodes
Description: Clinical interventions used to manage episodes of serious rash in participants could include topical corticosteroid (TC), intravenous (IV) and/or oral (PO) corticosteroids (IV/PO CS), emollients/moisturizers (E/M), antihistamines (AH), other treatment (OT), and CHC treatment regimen modifications including drug dose reduction (DDR), drug discontinuation (DD), and drug interruption (DI). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive).
  For each CHC treatment exposure group, the percentage of serious rash episodes managed by a particular intervention are reported out of the total number of managed serious rash episodes with data available for that intervention (i.e. serious rash episodes with missing data for an intervention were excluded).
Time Frame: Up to 48 weeks of a treatment regimen
Population: as for outcome 14
Measure: Number; unit: percentage of episodes
Units Other Than Participants: managed serious rash episodes total
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure
Number analyzed (Participants) | 1 | 7 | 26
Number analyzed (managed serious rash episodes total) | 1 | 7 | 26
percentage of episodes
  TC (managed episodes =1, 7, 26) | 100.0 [2.5 to 100.0] | 42.9 [59.0 to 100.0] | 65.4 [81.0 to 99.9]
  IV/PO CS (managed episodes =1, 7, 26) | 0.0 [0.0 to 97.5] | 28.6 [0.0 to 41.0] | 23.1 [0.1 to 19.0]
  E/M (managed episodes =1, 7, 26) | 100.0 | 28.6 | 23.1
  AH (managed episodes =1, 7, 26) | 100.0 | 28.6 | 73.1
  OT (managed episodes =1, 7, 26) | 0.0 | 14.3 | 15.4
  DDR (managed episodes =1, 3, 17) | 0.0 | 0.0 | 11.8
  DD (managed episodes =1, 3, 17) | 100.0 | 100.0 | 88.2
  DI (managed episodes =1, 3, 17) | 0.0 | 0.0 | 29.4

16. Secondary Outcome: Incidence of Anemia, Grade 3/4 Neutropenia, Grade 3/4 Thrombocytopenia, and Serious Skin Rash
Description: The incidence (events per 1000 participant-days) of the protocol-defined HOIs (anemia, grade 3/4 neutropenia, grade 3/4 thrombocytopenia, and serious skin rash) was calculated over the 48-week period following the start of CHC treatment exposure. All protocol-defined HOIs were taken into account (serious and non-serious HOIs). For this analysis, participants were categorized by CHC treatment group of exposure, and could successively be assigned to different treatment groups of exposure depending on their treatment regimen (treatment groups were not mutually exclusive). The incidence per 1000 participant-days of anemia, grade 3/4 neutropenia, grade 3/4 thrombocytopenia, and serious skin rash were reported by CHC treatment group of exposure with 95% confidence intervals.
Time Frame: Up to 48 weeks of treatment
Population: Participants in Analysis Population (CHC genotype-1 participants meeting eligibility criteria and treated with boceprevir+PR, telaprevir+PR, or PR alone) with available data who did not already experience HOI during 3 months preceding CHC treatment regimen. Participants categorized by treatment group of exposure further described in Arm Description
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-days
Arm/Group | PR Group of Exposure | Boceprevir + PR Group of Exposure | Telaprevir + PR Group of Exposure | PR + Boceprevir + Telaprevir Group of Exposure
Number analyzed (Participants) | 394 | 298 | 307 | 6
events per 1000 participant-days
  Anemia (n=391, 296, 306, 6) | 1.185 [0.767 to 1.749] | 3.302 [2.760 to 3.918] | 3.001 [2.499 to 3.572] | 5.122 [1.395 to 13.113]
  Grade 3/4 Neutropenia (n=394, 297, 307, 5) | 1.305 [0.860 to 1.899] | 1.656 [1.315 to 2.058] | 0.807 [0.591 to 1.077] | 3.195 [0.659 to 9.337]
  Grade 3/4 Thrombocytopenia (n=390, 295, 304, 6) | 0.835 [0.495 to 1.319] | 0.757 [0.544 to 1.027] | 0.596 [0.413 to 0.832] | 1.556 [0.188 to 5.622]
  Serious Rash (n=394, 298, 307, 6) | 0.045 [0.001 to 0.253] | 0.117 [0.047 to 0.242] | 0.430 [0.281 to 0.630] | 0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Up to 14 days following a 48-week treatment regimen (up to 50 weeks)
Description: AEs reported for Analysis Population by CHC treatment arms (mutually exclusive). Nonserious AEs (NSAEs) that were non-HOIs were not actively solicited on this study, however spontaneous drug-related NSAEs were collected and reported. As prespecified by the protocol, AEs were not collected for the PR Alone Arm until after amendment 3 (6/18/2013).
Arm/Group | Boceprevir + PR | Telaprevir + PR | PR Alone
Serious Adverse Events (participants affected / at risk) | 58/298 | 50/307 | 8/74
Other Adverse Events (participants affected / at risk) | 178/298 | 173/307 | 25/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir + PR (N=298) | Telaprevir + PR (N=307) | PR Alone (N=74)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 4 (4) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Long QT syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oral administration complication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative abscess (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Detoxification (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Liver transplant (Surgical and medical procedures) | 0 (0) | 3 (3) | 0 (0)
Oesophageal variceal ligation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Renal lithiasis prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Therapeutic embolisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir + PR (N=298) | Telaprevir + PR (N=307) | PR Alone (N=74)
Anaemia (Blood and lymphatic system disorders) | 133 (184) | 130 (173) | 9 (13)
Neutropenia (Blood and lymphatic system disorders) | 89 (130) | 49 (70) | 11 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 53 (67) | 37 (56) | 10 (15)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 30 (31) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a non-interventional study that collected data on both boceprevir and telaprevir treatment regimens within routine medical practice. No individual administration of any therapeutic or prophylactic agent was assigned in this protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.